CLINICAL TRIAL: NCT00254995
Title: Post-licensure Safety Surveillance Study of Routine Use of Meningococcal (Groups A, C, Y, and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine (Menactra ™)
Brief Title: Descriptive, Post-marketing, Surveillance Safety Study of Menactra Vaccine
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: MTA30
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Results first posted 2014-11-11 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Meningitis; Meningococcal Disease
Keywords: Meningitis; Meningococcal disease; Menactra vaccine
MeSH Terms: conditions — Meningitis; Meningococcal Infections

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Menactra Vaccine Recipients: Participants who received Menactra vaccine as part of routine medical care during the study period in Kaiser Permanente.
  Interventions: Biological: None administered in this study
- Age-Matched Control: Each individual receiving Menactra vaccine served as their own control for evaluation of acute (Days 0-30) events (short-term surveillance). For the 6-month (long-term) surveillance, for each person receiving Menactra vaccine, a control matched on age (± 1 year), sex, and month of vaccination was selected who received a received tetanus and diphtheria toxoids (Td), hepatitis A, hepatitis B, or hepatitis A/hepatitis B combination vaccine as part of routine medical care during the same month 1 year earlier in Kaiser Permanente
  Interventions: Biological: None administered in this study

INTERVENTIONS:
Biological: None administered in this study — N/A in this study

SUMMARY:
To further characterize the safety profile of Menactra vaccine and to identify any signals of potentially vaccine-related adverse events (AEs) not detected during pre-licensure studies.

ELIGIBILITY:
Inclusion Criteria:

* Receipt of Menactra vaccine during the study period.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Past receipt of Menactra vaccine
Sampling Method: Non-Probability Sample
Enrollment: 62626 (Actual)
Dates: Start 2005-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Oakland, California, United States

REFERENCES:
- [Derived] Hansen J, Zhang L, Klein NP, Robertson CA, Decker MD, Greenberg DP, Bassily E, Baxter R. Post-licensure safety surveillance study of routine use of quadrivalent meningococcal diphtheria toxoid conjugate vaccine. Vaccine. 2017 Dec 14;35(49 Pt B):6879-6884. doi: 10.1016/j.vaccine.2017.09.032. Epub 2017 Sep 21. PMID 28941623
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participant accrual occurred from 15 July 2005 through 14 April 2006.
Pre-assignment Details: Databases were reviewed to identify persons who received Menactra vaccine within Kaiser Permanente and to identify all medical care events for the 6-month period following vaccination or, if applicable, through the end of pregnancy. Subjects served as their own control for 0-30 days surveillance, age-matched control served for the 6-month period.
Groups:
- Menactra Vaccine Recipients: Kaiser Permanente members who received Menactra vaccine during the study period.
  Kaiser Permanente databases were used; Menactra vaccine was administered according to routine clinical practice.
- Control Group: Each individual receiving Menactra vaccine served as their own control for evaluation of acute (Days 0-30) events (short-term surveillance). For the 6-month (long-term) surveillance, for each person receiving Menactra vaccine, a control matched on age (± 1 year), sex, and month of vaccination was selected who received a received tetanus and diphtheria toxoids (Td), hepatitis A, hepatitis B, or hepatitis A/hepatitis B combination vaccine during the same month 1 year earlier.
  Kaiser Permanente databases were used; Menactra and control vaccine were administered according to routine clinical practice.
Period: Overall Study
Arm/Group | Menactra Vaccine Recipients | Control Group
Started | 31561 | 31065
Completed | 31561 | 31065
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects who received Menactra vaccine during the study period from the Kaiser Permanente databases.
Groups:
- Menactra Vaccine Recipients: Kaiser Permanente members who received Menactra vaccine during the study period.
  Kaiser Permanente database was used as no study vaccine was provided or administered as part of this study.
- Control Group: Each individual receiving Menactra vaccine served as their own control for evaluation of acute (Days 0-30) events (short-term surveillance). For the 6-month (long-term) surveillance, for each person receiving Menactra vaccine, a control matched on age (± 1 year), sex, and month of vaccination was selected who received a received tetanus and diphtheria toxoids (Td), hepatitis A, hepatitis B, or hepatitis A/hepatitis B combination vaccine during the same month 1 year earlier.
  Kaiser Permanente database was used as no study vaccine was provided or administered as part of this study.
- Total: Total of all reporting groups
Arm/Group | Menactra Vaccine Recipients | Control Group | Total
Number analyzed (Participants) | 31561 | 31065 | 62626
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.6 (5.56) | 15.65 (5.56) | 15.6 (5.56)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26805 | 26383 | 53188
  Between 18 and 65 years | 4732 | 4658 | 9390
  >=65 years | 24 | 24 | 48
Gender [Number; unit: Participants] — Gender information for 3 participants was not available in the database.
  Participants
    Female | 15722 | 15369 | 31091
    Male | 15836 | 15696 | 31532
Region of Enrollment [Number; unit: participants]
  United States | 31561 | 31065 | 62626
Seasonality [Number; unit: Participants] — Data represents participants receiving vaccine each season or time period shown. Some participants (49) had received more than one dose of Menactra vaccine are counted for each dose in the seasonality section.
  Participants
    December - February | 4689 | 4671 | 9360
    March - May | 3605 | 3602 | 7207
    June - August | 17577 | 17080 | 34657
    September - November | 5739 | 5712 | 11451

OUTCOME MEASURES:

1. Primary Outcome: Summary of Diagnoses With Significantly Elevated Findings From Risk-Window vs. Control-Window Comparisons: All Ages Combined - Short-Term Passive Surveillance
Description: Incidence rates for each diagnosis were calculated as the number of events divided by person-time and expressed as events per 1,000 person-months in each 30-day comparison window. Individuals receiving Menactra vaccine served as their own controls for evaluation of acute (Days 0-30) events. Rates of events occurring during Days 0-30 following vaccination were compared to rates of events occurring during Days 31-60 following vaccination. Clinical setting is given in parenthesis as either (H) for hospital or (ER) for emergency room.
Time Frame: Day 0 up to Day 60 post-vaccination
Population: All persons who received Menactra vaccine during the study period were included in the analysis.
Measure: Number; unit: Events per 1,000 person-months
Groups:
- Menactra Vaccine Recipients: Participants who received Menactra vaccine during the study period from the Kaiser Permanente databases.
  None administered in this study: N/A in this study
- Control Group: The individuals receiving Menactra vaccine served as their own controls for evaluation of acute (Days 0-30) events. Rates of events occurring during Days 0-30 following vaccination were compared to rates of events occurring during Days 31-60 following vaccination.
  The 6-month surveillance: For each individual receiving Menactra vaccine, a control matched on age (± 1 year), sex, and month of vaccination was selected who received a vaccination1 during the same month 1 year earlier. Rates of events occurring during the 6 months following vaccination with Menactra vaccine were compared to rates of events occurring during the 6 months following vaccination in the control individuals.
Arm/Group | Menactra Vaccine Recipients | Control Group
Number analyzed (Participants) | 31561 | 31065
Events per 1,000 person-months
  Abdominal pain (ER) | 0.98 | 0.52
  Febrile illness (ER) | 0.38 | 0.03
  Suicidal Ideation/Attempt (ER) | 0.19 | 0.00

2. Other Pre Specified Outcome: Summary of Diagnoses With Significantly Elevated Findings for Menactra Vaccine Recipients vs. Age-Matched Controls - All Ages Combined - Long-Term Passive Surveillance
Description: Incidence rates for each diagnosis were calculated as the number of events divided by person-time and expressed as events per 1,000 person-months in the 6-month surveillance period. For each individual receiving Menactra vaccine, a control matched on age (± 1 year), sex, and month of vaccination was selected who received a vaccination during the same month 1 year earlier. Rates of events occurring during the 6 months following vaccination with Menactra vaccine were compared to rates of events occurring during the 6 months following vaccination in age-matched controls. Clinical setting is given in parenthesis as either (H) for hospital or (ER) for emergency room.
Time Frame: Day 0 up to Day 180 post-vaccination
Population: All persons who received Menactra vaccine during the study period were included in the analysis.
Measure: Number; unit: Events per 1,000 person-months
Groups:
- Control Group: For each individual receiving Menactra vaccine, a control matched on age (± 1 year), sex, and month of vaccination was selected who received a vaccination1 during the same month 1 year earlier. Rates of events occurring during the 6 months following vaccination with Menactra vaccine were compared to rates of events occurring during the 6 months following vaccination in the control individuals.
Arm/Group | Menactra Vaccine Recipients | Control Group
Number analyzed (Participants) | 31561 | 31065
Events per 1,000 person-months
  Elective procedure (H) | 0.19 | 0.09
  Febrile illness (ER) | 0.25 | 0.13
  Genital pain (ER) | 0.03 | 0.00
  Hyperglycemia (ER) | 0.03 | 0.00
  Mononucleosis (ER) | 0.03 | 0.00
  Tympanic perforation (H) | 0.03 | 0.00
  Vomiting (ER) | 0.21 | 0.11

3. Other Pre Specified Outcome: Summary of Diagnoses With Significantly Elevated Findings From Risk-Window vs. Control-Window Comparisons - By Age Categories - Short-Term Passive Surveillance
Description: Incidence rates for each diagnosis were calculated as the number of events divided by person-time and expressed as events per 1,000 person-months for each 30-day comparison window. Individuals receiving Menactra vaccine served as their own controls for evaluation of acute (Days 0-30) events. Rates of events occurring during Days 0-30 following vaccination were compared to rates of events occurring during Days 31-60 following vaccination. Clinical setting is given in parenthesis as either (H) for hospital or (ER) for emergency room.
Time Frame: Day 0 up to Day 60 post-vaccination
Population: All persons who received Menactra vaccine during the study period were included in the analysis.
Measure: Number; unit: Events per 1,000 person-months
Groups:
- Control Group: Individuals receiving Menactra vaccine served as their own controls for evaluation of acute (Days 0-30) events. Rates of events occurring during Days 0-30 following vaccination were compared to rates of events occurring during Days 31-60 following vaccination.
Arm/Group | Menactra Vaccine Recipients | Control Group
Number analyzed (Participants) | 21407 | 21407
Events per 1,000 person-months
  Adominal pain (age 11-16 years; ER) | 1.07 | 0.38
  Febrile illness (age 11-16 years; ER) | 0.33 | 0.05
  Suicidal Ideation/Attempt (age 11-16 years; ER) | 0.23 | 0.00

4. Other Pre Specified Outcome: Summary of Diagnoses With Significantly Elevated Findings for Menactra Vaccine Recipients vs. Age-Matched Controls - By Age Categories - Long-Term Passive Surveillance
Description: Incidence rates for each diagnosis were calculated as the number of events divided by person-time and expressed as events per 1,000 person-months in the 6-month surveillance period. For each individual receiving Menactra vaccine, a control matched on age (± 1 year), sex, and month of vaccination was selected who received a vaccination during the same month 1 year earlier. Rates of events occurring during the 6 months following vaccination with Menactra vaccine were compared to rates of events occurring during the 6 months following vaccination in age-matched controls. Clinical setting is given in parenthesis as (C) for pre-specified adverse events, (H) for hospital, (ER) for emergency room.
Time Frame: Day 0 up to Day 180 post-vaccination
Population: All persons who received Menactra vaccine and their age-matched controls during the study period were included in the analysis.
Measure: Number; unit: Events per 1,000 person-months
Arm/Group | Menactra Vaccine Recipients | Control Group
Number analyzed (Participants) | 21407 | 21407
Events per 1,000 person-months
  Diabetes Type 1 (Prior onset)[age 11-16 years; ER] | 0.04 | 0.00
  Difficulty breathing/SOB (age 11-16 years; ER) | 0.07 | 0.02
  Elective procedure (age 11-16 years; H) | 0.20 | 0.06
  Febrile illness (age 11-16 years; ER) | 0.23 | 0.12
  Hives/Urticaria (age 11-16 years; C) | 0.40 | 0.24
  Mononucleosis (age 17-18 years; ER) | 0.10 | 0.00
  Otitis Externa (age 11-16 years; ER) | 0.04 | 0.00
  Vomiting (age 11-16 years; ER) | 0.18 | 0.09

5. Other Pre Specified Outcome: Summary of Diagnoses With Significantly Reduced Findings for Menactra Vaccine Recipients vs. Age-Matched Controls - All Ages Combined - Long-Term Passive Surveillance
Description: as for outcome 2
Time Frame: Day 0 up to Day 180 post-vaccination
Population: All persons who received Menactra vaccine during the study period were included in the analysis.
Measure: Number; unit: Events per 1,000 person-months
Arm/Group | Menactra Vaccine Recipients | Control Group
Number analyzed (Participants) | 31561 | 31065
Events per 1,000 person-months
  Abscess/Cellulitis (ER) | 0.12 | 0.25
  Allergic reaction (ER) | 0.01 | 0.06
  Allergy, drug (ER) | 0.00 | 0.03
  Benign lesion (H) | 0.12 | 0.24
  Congenital anomaly (H) | 0.10 | 0.18
  Cyst (H) | 0.04 | 0.10
  Fatigue (ER) | 0.01 | 0.04
  Insect bite (ER) | 0.01 | 0.05
  Musculoskeletal pain (ER) | 0.27 | 0.39
  Pelvic pain (ER) | 0.01 | 0.08
  Poisoning/Ingestion (H) | 0.02 | 0.07
  Post-operative complication (ER) | 0.01 | 0.07
  Post-operative complication (H) | 0.01 | 0.04
  Pregnancy delivery (H) | 0.00 | 0.03
  Psychiatric (ER) | 0.44 | 0.70
  Psychiatric (H) | 0.33 | 0.58
  Testicular pain (ER) | 0.01 | 0.05
  Tonsillitis (H) | 0.09 | 0.28
  Trauma (ER) | 3.77 | 5.13
  Vision disorder (H) | 0.01 | 0.05
  Well care/Reassurance/Follow-up (ER) | 0.07 | 0.24

6. Other Pre Specified Outcome: Summary of Diagnoses With Significantly Reduced Findings for Menactra Vaccine Recipients vs. Age-Matched Controls - By Age Categories - Long-Term Passive Surveillance
Description: as for outcome 2
Time Frame: Day 0 up to Day 180 post-vaccination
Population: All persons who received Menactra vaccine during the study period were included in the analysis.
Measure: Number; unit: Events per 1,000 person-months
Arm/Group | Menactra Vaccine Recipients | Control Group
Number analyzed (Participants) | 31392 | 31065
Events per 1,000 person-months
  Abdominal pain (age 30-55 years; ER) | 0.21 | 1.89
  Abscess/Cellulitis (age 11-16 years; ER) | 0.06 | 0.13
  Allergic reaction (age 11-16 years; ER) | 0.00 | 0.04
  Benign lesion (age 11-16 years; H) | 0.09 | 0.22
  Congenital anomaly (age 11-16 years; H) | 0.09 | 0.21
  Cyst (age 11-16 years; H) | 0.03 | 0.09
  Pelvic pain (age 17-18 years; ER) | 0.00 | 0.17
  Post-operative complication (age 17-18 years; ER) | 0.02 | 0.15
  Psychiatric (age 11-16 years; H) | 0.32 | 0.52
  Psychiatric (age 17-18 years; ER) | 0.43 | 1.34
  Psychiatric (age 17-18 years; H) | 0.38 | 0.77
  Testicular pain (age 11-16 years; ER) | 0.01 | 0.06
  Tonsillitis (age 11-16 years; H) | 0.09 | 0.26
  Tonsillitis (age 17-18 years; ER) | 0.04 | 0.22
  Tonsillitis (age 17-18 years; H) | 0.10 | 0.39
  Trauma (age 11-16 years; ER) | 3.88 | 4.66
  Trauma (age 17-18 years; ER) | 3.62 | 5.27
  Trauma (age 19-29 years; ER) | 3.53 | 10.9
  Trauma (age 19-29 years; H) | 0.00 | 1.28
  Trauma (age 30-55 years; ER) | 2.52 | 9.41
  Trauma (age 30-55 years; H) | 0.00 | 1.05
  Well care/Reassurance/Follow-up (age 11-16 yrs;ER) | 0.05 | 0.17
  Well care/Reassurance/Follow-up (age 17-18 yrs;ER) | 0.10 | 0.37

7. Other Pre Specified Outcome: Rates of Serious Adverse Events Per 1000 Doses During 6 Months After Menactra Vaccination - ER Setting - All Ages Combined.
Description: Only persons who received Menactra vaccine during the study period were surveyed and included in this outcome.
Time Frame: Day 0 up to 6 months post-vaccination
Population: Only all persons who received Menactra vaccine during the study period were included in the analysis.
Measure: Number; unit: Events per 1,000 doses
Groups:
- Control Group: The 6-month surveillance: For each individual receiving Menactra vaccine, a control matched on age (± 1 year), sex, and month of vaccination was selected who received a vaccination1 during the same month 1 year earlier. Rates of events occurring during the 6 months following vaccination with Menactra vaccine were compared to rates of events occurring during the 6 months following vaccination in the control individuals.
Arm/Group | Menactra Vaccine Recipients | Control Group
Number analyzed (Participants) | 31561 | 0
Events per 1,000 doses
  Cardiac arrest | 0.03 |
  Pregnancy | 0.03 |

8. Other Pre Specified Outcome: Rates of Serious Adverse Events Per 1000 Doses at During 6 Months After Menactra Vaccination - Hospital Setting - All Ages Combined
Description: Only persons who received Menactra vaccine during the study period were surveyed and included in this outcome.
Time Frame: Day 0 up to 6 months post-vaccination
Population: Only persons who received Menactra vaccine during the study period were included in the analysis.
Measure: Number; unit: Events per 1,000 doses
Arm/Group | Menactra Vaccine Recipients | Control Group
Number analyzed (Participants) | 31561 | 0
Events per 1,000 doses
  Abdominal pain | 0.06 |
  Abscess/Cellulitis | 0.38 |
  Acute renal failure | 0.03 |
  Appendicitis | 0.57 |
  Arrhythmia | 0.03 |
  Aseptic meningitis | 0.03 |
  Asphyxiation | 0.03 |
  Asthma/Reactive airway disease | 0.16 |
  Benign lesion | 0.16 |
  COPD | 0.03 |
  Cancer, Cervix | 0.03 |
  Cancer, Melanoma | 0.03 |
  Cancer, Ovarian | 0.03 |
  Cancer, Pancreatic | 0.03 |
  Cancer, Rule out cancer | 0.16 |
  Cholelithiasis | 0.06 |
  Chronic inflammatory demyelinating polyneuritis | 0.03 |
  Complications of transplanted organ | 0.03 |
  Congenital anomaly | 0.38 |
  Congenital heart disease | 0.03 |
  Constipation | 0.06 |
  Cranial nerve palsy | 0.03 |
  Cyst | 0.13 |
  Dehydration | 0.10 |
  Delirium tremens | 0.03 |
  Dental | 0.10 |
  Diabetes type I (Diagnosed after vaccination) | 0.10 |
  Diabetes type I (Diagnosed before vaccination) | 0.13 |
  Diarrhea | 0.03 |
  Elective procedure | 0.22 |
  Encephalitis | 0.03 |
  Encephalitis due to Epstein-Barr virus | 0.03 |
  End-stage renal disease | 0.03 |
  Epilepsy (Hx of seizure disorder possible seizure) | 0.03 |
  Epilepsy (Seizure event, w/hx of seizure disorder) | 0.06 |
  Fatty liver | 0.03 |
  Febrile illness | 0.06 |
  Femoral epiphysiolysis | 0.03 |
  Foreign body | 0.03 |
  Gastroesophageal reflux | 0.03 |
  Gastroenteritis | 0.19 |
  Hodgkin's disease | 0.03 |
  Horner's syndrome | 0.03 |
  Hydrocephalus | 0.03 |
  Hypertension | 0.03 |
  ITP (Diagnosed before vaccination) | 0.06 |
  Idiopathic polycystic splenomegaly | 0.03 |
  Inguinal hernia/repair | 0.03 |
  Kyphosis | 0.03 |
  Labyrinthitis | 0.03 |
  Lymphocytic leukemia (Chronic, diagnosed before) | 0.03 |
  Migraine | 0.06 |
  Osteomyelitis | 0.03 |
  Pancreatitis | 0.03 |
  Pectus excavatum | 0.03 |
  Pelvic inflammatory disease | 0.03 |
  Pharyngitis | 0.03 |
  Pneumocystosis | 0.03 |
  Pneumonia | 0.13 |
  Pneumothorax | 0.03 |
  Poisoning/ingestion | 0.06 |
  Pregnancy | 0.03 |
  Pregnancy - Stillborn delivery post prolapsed cord | 0.03 |
  Psychiatric | 1.93 |
  Plumonary embolism | 0.03 |
  Respiratory syncytial virus infection | 0.03 |
  Renal calculus | 0.03 |
  Scoliosis | 0.19 |
  Sickle cell disease | 0.10 |
  Sleep apnea | 0.03 |
  Splenomegaly | 0.03 |
  Suicidal ideation/attempt | 0.03 |
  Syncope/Loss of consciousness | 0.10 |
  SLE (Diagnosed after vaccination; symptoms before) | 0.03 |
  SLE (Diagnosed before vaccination) | 0.03 |
  Temporomandibular joint disorder | 0.19 |
  Testicular torsion | 0.03 |
  Thrombocytopenia (Chronic, diagnosed before vacc.) | 0.10 |
  Tonsillitis | 0.03 |
  Toxic shock syndrome | 0.03 |
  Transplant rejection | 0.03 |
  Trauma | 1.20 |
  Urinary tract infection | 0.10 |
  Viral syndrome | 0.03 |

9. Other Pre Specified Outcome: Summary of Reported Pregnancy Outcomes in Menactra Vaccine Recipients Pregnant at or Within 28 Days After Vaccination
Description: Only persons who received Menactra vaccine during the study period were included in this outcome.
Time Frame: Day 0 up to Determination of Pregnancy Outcome
Population: Only persons who received Menactra vaccine during the study period were included in the analysis. There were no control group analysis because the threshold of 25 pregnancies with known were not achieved at the time the surveillance was concluded.
Measure: Number; unit: Paticipants
Arm/Group | Menactra Vaccine Recipients | Control Group
Number analyzed (Participants) | 31561 | 0
Paticipants
  Live births | 11 |
  Live births with congenital anomaly (facial cyst) | 1 |
  Elective abortion | 5 |
  Early fetal death | 1 |
  Lost to follow up | 7 |

ADVERSE EVENTS:
Time Frame: Adverse events data surveillance period was from the day of vaccination up to 6 months post-vaccination from the Hospital database.
Arm/Group | Menactra Vaccine Recipients
Serious Adverse Events (participants affected / at risk) | 273/31561
Other Adverse Events (participants affected / at risk) | 0/31558
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Menactra Vaccine Recipients (N=31561)
Thrombocytopenia (Chronic, Precedes) (Blood and lymphatic system disorders) | 3
Idiopathic thrombocytopenic purpura (Precedes) (Blood and lymphatic system disorders) | 2
Splenomegaly (Blood and lymphatic system disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Congenital Anomaly (Congenital, familial and genetic disorders) | 12
Congenital Heart Disease (Congenital, familial and genetic disorders) | 1
Sickle Cell Disease (Congenital, familial and genetic disorders) | 3
Pectus Excavatum (Congenital, familial and genetic disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Gastrooesophageal reflux (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Cyst (General disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 3
Febrile Illness (General disorders) | 2
Delirium Tremens (Psychiatric disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Fatty Liver (Hepatobiliary disorders) | 1
Transplant Rejection (Immune system disorders) | 1
Abscess/Cellulitis (Infections and infestations) | 12
Appendicitis (Infections and infestations) | 18
Gastroenteritis (Infections and infestations) | 6
Pneumonia (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 3
Aseptic Meningitis (Infections and infestations) | 1
Encephalitis due to Epstein-Barr Virus (Infections and infestations) | 1
Viral Syndrome (Infections and infestations) | 1
Pelvic Inflammatory Disease (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Labyrinthitis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Toxic Shock Syndrome (Infections and infestations) | 1
Complications of Transplanted Organ (Injury, poisoning and procedural complications) | 1
Foreign Body (Injury, poisoning and procedural complications) | 1
Poisoning/Ingestion (Injury, poisoning and procedural complications) | 2
Trauma (Injury, poisoning and procedural complications) | 38
Diabetes, Type 1 (New Onset) (Metabolism and nutrition disorders) | 3
Diabetes, Type 1 (Prior Onset) (Metabolism and nutrition disorders) | 4
Femoral Epiphysiolysis (Musculoskeletal and connective tissue disorders) | 1
Kyphosis (Musculoskeletal and connective tissue disorders) | 1
Systemic Lupus Erythematosus (New dx, symptoms precede) (Musculoskeletal and connective tissue disorders) | 1
Systemic Lupus Erythematosus (Prior onset) (Musculoskeletal and connective tissue disorders) | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 6
Temporomandibular Joint Disorder (Musculoskeletal and connective tissue disorders) | 6
Cancer, Cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cancer, Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cancer, Ovarian (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cancer, Pancreatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign lesion NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Cancer, R/O Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphocytic Leukemia (Chronic, Precedes) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Encephalitis (Nervous system disorders) | 1
Cranial Nerve Palsy (Nervous system disorders) | 1
Chronic Inflammatory Demyelinating Polyneuritis (Prior onset) (Nervous system disorders) | 1
Epilepsy (Hx of Seizure Disorder, possible seizure) (Nervous system disorders) | 1
Epilepsy (Seizure Event, w/hx of Seizure Disorder) (Nervous system disorders) | 2
Horner's Syndrome (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 2
Syncope/LOC (Nervous system disorders) | 3
Pregnancy (Reproductive system and breast disorders) | 1
Pregnancy - Stillborn Delivery post Prolapsed Cord (Reproductive system and breast disorders) | 1
Psychiatric (Psychiatric disorders) | 61
Suicidal Ideation/Attempt (Psychiatric disorders) | 1
Acute Renal Failure (Renal and urinary disorders) | 1
Renal Calculus (Renal and urinary disorders) | 1
End-Stage Renal Disease (Renal and urinary disorders) | 1
Testicular Torsion (Reproductive system and breast disorders) | 1
Asthma/RAD (Respiratory, thoracic and mediastinal disorders) | 5
Asphyxiation (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 1
Elective Procedure (Surgical and medical procedures) | 7
Inguinal Hernia/Repair (Surgical and medical procedures) | 1
Tooth disorder (Dental) (Gastrointestinal disorders) | 3
Hypertension (Vascular disorders) | 1
Idiopathic Polycystic Splenomegaly (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pneumocystosis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.